CLINICAL TRIAL: NCT03426709
Title: Efficacy of a Blended Low Intensity Internet-delivered Psychological Program in Patients With Multimorbidity in Primary Care. A Randomized Clinical Trial.
Brief Title: Efficacy of a Blended Low Intensity Internet-delivered Psychological Program in Patients With Multimorbidity in Primary Care.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Javier Garcia Campayo (Other)
Collaborators: Carlos III Health Institute (Other Government)
Responsible Party: Sponsor-Investigator, Javier Garcia Campayo, Principal investigator, Hospital Miguel Servet
Organization: Hospital Miguel Servet (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PI16/00962
Record Dates: First submitted 2018-02-02; First posted 2018-02-08 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Depression; Chronic Disease (Diabetes/Low Back Pain)
Keywords: Depression; Multimorbidity; Computer-delivered psychotherapy; Randomized-controlled trial; Cost-effectiveness
MeSH Terms: conditions — Depression; Chronic Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low intensity Internet-delivered psychotherapy (Experimental): improved Treatment-as-usual (TAU) + face to face (2 sessions of 90 minutes/session) + low intensity psychological intervention (6 sessions of 60 minutes/session) applied by ICTs (Information and communication technologies).
  Interventions: Behavioral: Low intensity Internet-delivered psychotherapy
- Improved Treatment-as-usual (TAU) (No Intervention): In this group, the general practitioner (GP) will apply the usual but improved treatment. The GP will have a training meeting and will be provided with the recommendations of one of the Guidelines for the Treatment of Adult Depression in AP most used in our country.

INTERVENTIONS:
Behavioral: Low intensity Internet-delivered psychotherapy — The online intervention will be individual and interactive, which will be supported by multimedia material (videos, sound recordings, etc.) and will have internet support. The estimated duration of the program is 8 weeks. Low Intensity Internet-delivered psychotherapy: Psychoeducation, Healthy living habits, Behavioral activation, Positive Psychology, Mindfulness and Compassion
  Arms: Low intensity Internet-delivered psychotherapy

SUMMARY:
The aim of this study is to assess the efficacy in Primary Care (PC) of a low intensity psychological intervention applied using Information and communication technologies (ICTs) for the treatment of multimorbidity in PC (depression and diabetes/low back pain) by a randomized controlled trial (RCT). A protocol will be design that combines face to face intervention with a supporting online program that will be tried in a RCT conducted in 3 different regions (Andalucía, Aragón, y Baleares). Our main hypothesis is that improved usual care combined with psychological therapy applied by ICTs, will be more efficacious to improve the symptomatology of multimorbidity, compared to a group with only improved treatment as usual three months after the end of treatment.

DETAILED DESCRIPTION:
Although multimorbidity is highly prevalent, health care systems are designed for the management individual diseases. New strategies are needed to help general practitioners to provide appropriate personalized care to patients. The World Health Organization (WHO) has included comorbidity between depression and a chronic disease as one of the 10 main priorities in global public health. Studies in meta-analysis confirm that the 2 main interventions of first choice for depression are pharmacotherapy and/or psychotherapy, with similar results in the short term but superior in the long term for psychological treatments. Given the difficulty of delivering face to face psychological treatments (high costs) alternative models of delivering treatments have been proposed, emphasizing the role of technologies like Internet. The aim of this study is to assess the efficacy in Primary Care (PC) of a low intensity psychological intervention (8 weeks) applied using Information and communication technologies (ICTs) for the treatment of multimorbidity in PC (depression and diabetes/low back pain) by a randomized controlled trial (RCT). Our main hypothesis is that improved usual care combined with psychological therapy applied by ICTs, will be more efficacious to improve the symptomatology of multimorbidity, compared to a group with only improved treatment as usual three months after the end of treatment. A protocol will be design that combines face to face intervention with a supporting online program that will be tried in a RCT conducted in 3 different regions (Andalucía, Aragón, y Baleares). 180 participants diagnosed with depression and diabetes/low back pain will participate in the RCT. It´s proposed a coordinated study by 4 highly experienced groups with great possibilities of translation and transference to usual clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Be adult
* Willingness to participate in the study and signing informed consent
* Ability to understand oral and written Spanish.
* DSM-5 diagnose of Major Depression or Dysthymia, mild or moderate depression expressed as score lower than 19 in the Patient Health Questionnaire (PHQ-9)
* Duration of depressive symptoms 2 months or more
* Diagnosis of one of the following two conditions: Diabetes (Diagnosis according to criteria of the American Diabetes Association (ADA)) or low back pain (Diagnosis of non-specific chronic low back pain according to the definition established by the Clinical Practice Guide of the European Program COST B-13 (CPG COST B-13) with a duration of at least 6 months)
* To have and to handle the computer, internet and mobile phone

Exclusion Criteria:

* Any diagnose of disease that may affect central nervous system (brain pathology, traumatic brain injury, dementia, etc.),
* Other psychiatric diagnoses or acute psychiatric illness (substance dependence or abuse, history of schizophrenia or other psychotic disorders, eating disorders, etc.), except for anxious pathology or personality disorders
* Any medical, infectious or degenerative disease that may affect mood
* Presence of delusional ideas or hallucinations consistent or not with mood
* Suicide risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | Baseline
  In the Intervention group. The Patient Health Questionnaire (PHQ-9) is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. PHQ scores ≥ 10 had a sensitivity of 88% and a specificity of 88% for major depression. PHQ-9 scores of 5, 10, 15, and 20 represents mild, moderate, moderately severe and severe depression. The possible range is 0-27.
Patient Health Questionnaire (PHQ-9) | Baseline
  In the TAU control group. The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. PHQ scores ≥ 10 had a sensitivity of 88% and a specificity of 88% for major depression. PHQ-9 scores of 5, 10, 15, and 20 represents mild, moderate, moderately severe and severe depression. The possible range is 0-27.
Patient Health Questionnaire (PHQ-9) | Post-treatment 8-12 weeks from baseline in the intervention group
  The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. PHQ scores ≥ 10 had a sensitivity of 88% and a specificity of 88% for major depression. PHQ-9 scores of 5, 10, 15, and 20 represents mild, moderate, moderately severe and severe depression. The possible range is 0-27.
Patient Health Questionnaire (PHQ-9) | Post-treatment 8-12 weeks from baseline in the TAU control group
  The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. PHQ scores ≥ 10 had a sensitivity of 88% and a specificity of 88% for major depression. PHQ-9 scores of 5, 10, 15, and 20 represents mild, moderate, moderately severe and severe depression. The possible range is 0-27.
Patient Health Questionnaire (PHQ-9) | 3 months follow up in the intervention group
  The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. PHQ scores ≥ 10 had a sensitivity of 88% and a specificity of 88% for major depression. PHQ-9 scores of 5, 10, 15, and 20 represents mild, moderate, moderately severe and severe depression. The possible range is 0-27.
Patient Health Questionnaire (PHQ-9) | 3 months follow up in the TAU control group
  The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. PHQ scores ≥ 10 had a sensitivity of 88% and a specificity of 88% for major depression. PHQ-9 scores of 5, 10, 15, and 20 represents mild, moderate, moderately severe and severe depression. The possible range is 0-27.
Patient Health Questionnaire (PHQ-9) | Every week, after the completion of the corresponding module, until the end of the intervention (for an average of 2 months).
  The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. PHQ scores ≥ 10 had a sensitivity of 88% and a specificity of 88% for major depression. PHQ-9 scores of 5, 10, 15, and 20 represents mild, moderate, moderately severe and severe depression. The possible range is 0-27.
Visual Analog Scale (0-100) or Numeric Pain Scale (0-10) | Baseline
  In the Intervention group
Visual Analog Scale (0-100) or Numeric Pain Scale (0-10) | Baseline
  In the TAU control group
Visual Analog Scale (0-100) or Numeric Pain Scale (0-10) | Post-treatment 8-12 weeks from baseline in the intervention group
Visual Analog Scale (0-100) or Numeric Pain Scale (0-10) | Post-treatment 8-12 weeks from baseline in the TAU control group
Visual Analog Scale (0-100) or Numeric Pain Scale (0-10) | 3 months follow up in the intervention group
Visual Analog Scale (0-100) or Numeric Pain Scale (0-10) | 3 months follow up in the TAU control group
Roland Morris Disability Questionnaire (RMDQ) | Baseline
  In the Intervention group. The Roland Morris Disability Questionnaire (RMDQ) consists of 24 statements relating to the person's perceptions of their back pain and associated disability. This includes items on physical ability/ activity (15), sleep/rest (3), psychosocial (2), household management (2), eating (1) and pain frequency (1). It is designed to take approximately 5 minutes to complete, without any assistance from the administrator. The RMDQ is scored by adding up the number of items checked by the patient (1 if is checked, 0 if is not). The score can range from 0 (no disability) to 24 (maximal disability).
Roland Morris Disability Questionnaire (RMDQ) | Baseline
  In the TAU control group. The Roland Morris Disability Questionnaire (RMDQ) consists of 24 statements relating to the person's perceptions of their back pain and associated disability. This includes items on physical ability/ activity (15), sleep/rest (3), psychosocial (2), household management (2), eating (1) and pain frequency (1). It is designed to take approximately 5 minutes to complete, without any assistance from the administrator. The RMDQ is scored by adding up the number of items checked by the patient (1 if is checked, 0 if is not). The score can range from 0 (no disability) to 24 (maximal disability).
Roland Morris Disability Questionnaire (RMDQ) | Post-treatment 8-12 weeks from baseline in the intervention group
  The Roland Morris Disability Questionnaire (RMDQ) consists of 24 statements relating to the person's perceptions of their back pain and associated disability. This includes items on physical ability/ activity (15), sleep/rest (3), psychosocial (2), household management (2), eating (1) and pain frequency (1). It is designed to take approximately 5 minutes to complete, without any assistance from the administrator. The RMDQ is scored by adding up the number of items checked by the patient (1 if is checked, 0 if is not). The score can range from 0 (no disability) to 24 (maximal disability).
Roland Morris Disability Questionnaire (RMDQ) | Post-treatment 8-12 weeks from baseline in the TAU control group
  The Roland Morris Disability Questionnaire (RMDQ) consists of 24 statements relating to the person's perceptions of their back pain and associated disability. This includes items on physical ability/ activity (15), sleep/rest (3), psychosocial (2), household management (2), eating (1) and pain frequency (1). It is designed to take approximately 5 minutes to complete, without any assistance from the administrator. The RMDQ is scored by adding up the number of items checked by the patient (1 if is checked, 0 if is not). The score can range from 0 (no disability) to 24 (maximal disability).
Roland Morris Disability Questionnaire (RMDQ) | 3 months follow up in the intervention group
  The Roland Morris Disability Questionnaire (RMDQ) consists of 24 statements relating to the person's perceptions of their back pain and associated disability. This includes items on physical ability/ activity (15), sleep/rest (3), psychosocial (2), household management (2), eating (1) and pain frequency (1). It is designed to take approximately 5 minutes to complete, without any assistance from the administrator. The RMDQ is scored by adding up the number of items checked by the patient (1 if is checked, 0 if is not). The score can range from 0 (no disability) to 24 (maximal disability).
Roland Morris Disability Questionnaire (RMDQ) | 3 months follow up in the TAU control group
  The Roland Morris Disability Questionnaire (RMDQ) consists of 24 statements relating to the person's perceptions of their back pain and associated disability. This includes items on physical ability/ activity (15), sleep/rest (3), psychosocial (2), household management (2), eating (1) and pain frequency (1). It is designed to take approximately 5 minutes to complete, without any assistance from the administrator. The RMDQ is scored by adding up the number of items checked by the patient (1 if is checked, 0 if is not). The score can range from 0 (no disability) to 24 (maximal disability).
Diabetes control measured by VR d= Hb glucosidal | Baseline
  In the Intervention group
Diabetes control measured by VR d= Hb glucosidal | Baseline
  In the TAU control group
Diabetes control measured by VR d= Hb glucosidal | Post-treatment 8-12 weeks from baseline in the intervention group
Diabetes control measured by VR d= Hb glucosidal | Post-treatment 8-12 weeks from baseline in the TAU control group
Diabetes control measured by VR d= Hb glucosidal | 3 months follow up in the intervention group
Diabetes control measured by VR d= Hb glucosidal | 3 months follow up in the TAU control group

SECONDARY OUTCOMES:
Sociodemographic data Gender, age, marital status, education, occupation, economical level | Baseline
  In the Intervention group and the TAU control group
The Mini-International Neuropsychiatric Interview (MINI) | Baseline
  In the Intervention group and the TAU control group. This is a short structured diagnostic psychiatric interview that yields key DSM-IV and ICD-10 diagnoses. MINI can be administered in a short period of time and clinical interviewers need only a brief training. The MINI has been translated and validated in Spanish.
Health Survey 12 (SF-12) | Baseline
  In the Intervention group
Health Survey 12 (SF-12) | Baseline
  In the TAU control group
Health Survey 12 (SF-12) | Post-treatment 12 weeks from baseline in the intervention group
Health Survey 12 (SF-12) | Post-treatment 12 weeks from baseline in the TAU control group
Health Survey 12 (SF-12) | 3 months follow up in the intervention group
Health Survey 12 (SF-12) | 3 months follow up in the TAU control group
Client Service Receipt Inventory (CSRI) | Baseline
  In the Intervention group
Client Service Receipt Inventory (CSRI) | Baseline
  In the TAU control group
Client Service Receipt Inventory (CSRI) | Post-treatment 12 weeks from baseline in the intervention group
Client Service Receipt Inventory (CSRI) | Post-treatment 12 weeks from baseline in the TAU control group
Client Service Receipt Inventory (CSRI) | 3 months follow up in the intervention group
Client Service Receipt Inventory (CSRI) | 3 months follow up in the TAU control group
Positive and Negative Affect Schedule (PANAS) | Baseline in the intervention group and TAU control group
  The PANAS is a self-report questionnaire that measure positive and negative affect and consists of a list of 20 adjectives (10 positive: e.g., "interested", and 10 negative: e.g., "guilty") that are rated on a 5-point Likert-type scale. This questionnaire has already been validated in the Spanish population with appropriate psychometric characteristics (Sandin et al., 1999).
Positive and Negative Affect Schedule (PANAS) | 3 months follow up in the intervention group and TAU control group
  The PANAS is a self-report questionnaire that measure positive and negative affect and consists of a list of 20 adjectives (10 positive: e.g., "interested", and 10 negative: e.g., "guilty") that are rated on a 5-point Likert-type scale. This questionnaire has already been validated in the Spanish population with appropriate psychometric characteristics (Sandin et al., 1999).
Positive and Negative Affect Schedule (PANAS) | Every week, after the completion of the corresponding module, until the end of the intervention (for an average of 2 months).
  The PANAS is a self-report questionnaire that measure positive and negative affect and consists of a list of 20 adjectives (10 positive: e.g., "interested", and 10 negative: e.g., "guilty") that are rated on a 5-point Likert-type scale. This questionnaire has already been validated in the Spanish population with appropriate psychometric characteristics (Sandin et al., 1999).
Positive and Negative Affect Schedule (PANAS) | Post-treatment 12 weeks from baseline in the intervention and TAU control group
  The PANAS is a self-report questionnaire that measure positive and negative affect and consists of a list of 20 adjectives (10 positive: e.g., "interested", and 10 negative: e.g., "guilty") that are rated on a 5-point Likert-type scale. This questionnaire has already been validated in the Spanish population with appropriate psychometric characteristics (Sandin et al., 1999).
Usefulness | Every week, after the completion of the corresponding module, until the end of the intervention (for an average of 2 months).
  A single question about usefulness (i.e., "To what extent has this module been useful to you?" (Lopez-Montoyo et al., 2019); with a Likert-type response option that ranges between 0 = "nothing" and 10 = "very much").
System Usability Scale (SUS) | Post module 1 (Psychoeducation) after an average of 1 week
  The SUS is a 10-item questionnaire that measures usability in relation to the quality and acceptability of the intervention (i.e., "I think that I would like to use this system frequently"; with a Likert-type response option that ranges between 1 = "strongly disagree" and 5 = "strongly agree") (Bangor et al., 2008).

CONTACTS AND LOCATIONS:
Overall Officials: Javier García-Campayo, Principal Investigator — Miguel Servet Hospital and University os Zaragoza, Spain
Locations (4):
- Spain (4):
  - Health Science Research Institute, University Balearic Islands, Palma de Mallorca, Mallorca
  - Psychiatric Service. University Hospital Carlos Haya, Málaga
  - Valencia University and CIBER Physiopathology of Obesity and Nutrition. Carlos III Health Institute, Valencia
  - Department of Psychiatry. Miguel Servet University Hospital, Zaragoza

REFERENCES:
- [Background] Bogner HR, de Vries HF. Integration of depression and hypertension treatment: a pilot, randomized controlled trial. Ann Fam Med. 2008 Jul-Aug;6(4):295-301. doi: 10.1370/afm.843. PMID 18626028
- [Background] Katon WJ, Lin EH, Von Korff M, Ciechanowski P, Ludman EJ, Young B, Peterson D, Rutter CM, McGregor M, McCulloch D. Collaborative care for patients with depression and chronic illnesses. N Engl J Med. 2010 Dec 30;363(27):2611-20. doi: 10.1056/NEJMoa1003955. PMID 21190455
- [Background] Andersson G, Cuijpers P. Internet-based and other computerized psychological treatments for adult depression: a meta-analysis. Cogn Behav Ther. 2009;38(4):196-205. doi: 10.1080/16506070903318960. PMID 20183695
- [Background] Kaltenthaler E, Parry G, Beverley C, Ferriter M. Computerised cognitive-behavioural therapy for depression: systematic review. Br J Psychiatry. 2008 Sep;193(3):181-4. doi: 10.1192/bjp.bp.106.025981. PMID 18757972
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Diez-Quevedo C, Rangil T, Sanchez-Planell L, Kroenke K, Spitzer RL. Validation and utility of the patient health questionnaire in diagnosing mental disorders in 1003 general hospital Spanish inpatients. Psychosom Med. 2001 Jul-Aug;63(4):679-86. doi: 10.1097/00006842-200107000-00021. PMID 11485122
- [Background] Ostelo RW, de Vet HC, Knol DL, van den Brandt PA. 24-item Roland-Morris Disability Questionnaire was preferred out of six functional status questionnaires for post-lumbar disc surgery. J Clin Epidemiol. 2004 Mar;57(3):268-76. doi: 10.1016/j.jclinepi.2003.09.005. PMID 15066687
- [Background] Stratford PW, Binkley J, Solomon P, Finch E, Gill C, Moreland J. Defining the minimum level of detectable change for the Roland-Morris questionnaire. Phys Ther. 1996 Apr;76(4):359-65; discussion 366-8. doi: 10.1093/ptj/76.4.359. PMID 8606899
- [Background] Kovacs FM, Llobera J, Gil Del Real MT, Abraira V, Gestoso M, Fernandez C, Primaria Group KA. Validation of the spanish version of the Roland-Morris questionnaire. Spine (Phila Pa 1976). 2002 Mar 1;27(5):538-42. doi: 10.1097/00007632-200203010-00016. PMID 11880841
- [Background] Gandek B, Ware JE, Aaronson NK, Apolone G, Bjorner JB, Brazier JE, Bullinger M, Kaasa S, Leplege A, Prieto L, Sullivan M. Cross-validation of item selection and scoring for the SF-12 Health Survey in nine countries: results from the IQOLA Project. International Quality of Life Assessment. J Clin Epidemiol. 1998 Nov;51(11):1171-8. doi: 10.1016/s0895-4356(98)00109-7. PMID 9817135
- [Background] Alonso J, Prieto L, Anto JM. [The Spanish version of the SF-36 Health Survey (the SF-36 health questionnaire): an instrument for measuring clinical results]. Med Clin (Barc). 1995 May 27;104(20):771-6. Spanish. PMID 7783470
- [Background] Ferrando L, Bobes J, Gilbert J, Soto M, Soto O. MINI: MINI International Neuropsychiatric Interview, Madrid, IAP, 1998.
- [Background] Beecham JK, et al. Costing psychiatric interventions. In: Thornicroft G, ed. Measuring mental health needs. London: Royal College of Psychiatrists; 2001; 200-224.
- [Background] Vazquez-Barquero JL. et al. Spanish version of the CSRI: a mental health cost evauation interview. Arch Neurobol, 1997; 60: 171-84.
- [Derived] Monreal-Bartolome A, Castro A, Perez-Ara MA, Gili M, Mayoral F, Hurtado MM, Varela Moreno E, Botella C, Garcia-Palacios A, Banos RM, Lopez-Del-Hoyo Y, Garcia-Campayo J, Montero-Marin J. Efficacy of a Blended Low-Intensity Internet-Delivered Psychological Program in Patients With Multimorbidity in Primary Care: Randomized Controlled Trial. J Med Internet Res. 2025 Feb 10;27:e56203. doi: 10.2196/56203. PMID 39928931
- [Derived] Varela-Moreno E, Anarte-Ortiz MT, Jodar-Sanchez F, Garcia-Palacios A, Monreal-Bartolome A, Gili M, Garcia-Campayo J, Mayoral-Cleries F. Economic Evaluation of a Web Application Implemented in Primary Care for the Treatment of Depression in Patients With Type 2 Diabetes Mellitus: Multicenter Randomized Controlled Trial. JMIR Mhealth Uhealth. 2024 May 16;12:e55483. doi: 10.2196/55483. PMID 38754101
- [Derived] Monreal-Bartolome A, Barcelo-Soler A, Castro A, Perez-Ara MA, Gili M, Mayoral F, Hurtado MM, Moreno EV, Botella C, Garcia-Palacios A, Banos RM, Lopez-Del-Hoyo Y, Garcia-Campayo J. Efficacy of a blended low-intensity internet-delivered psychological programme in patients with multimorbidity in primary care: study protocol for a randomized controlled trial. BMC Psychiatry. 2019 Feb 11;19(1):66. doi: 10.1186/s12888-019-2037-3. PMID 30744610
- See also: Official website of the Spanish Research Network in Primary Care (Rediapp) — http://www.rediapp.org/